CLINICAL TRIAL: NCT00637260
Title: Motor Cortex Stimulation for Parkinson's Disease. A Prospective Double Blind Randomized Study With Cross-over
Brief Title: Motor Cortex Stimulation for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University, Italy (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, bEATRICE CIONI, MD, Catholic University, Italy
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 820117
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Parkinson's Disease
Keywords: motorcortex stimulation; Parkinson's disease; neuromodulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Device: Motor cortex stimulation on.
- B (Sham Comparator)
  Interventions: Device: motor cortex stimulation off

INTERVENTIONS:
Device: Motor cortex stimulation on. — The parameters of stimulation will be: contact 0 cathode, contact 3anode, 120microsec, 80 Hz, subthreshold for any movement or sensation, usually 3-5Volts. The stimulator will be switched on, continuously.
  Other Names: Motor cortex stimulation on
  Arms: A
Device: motor cortex stimulation off — The parameters of stimulation will be: contact 0 cathode, contact 3 anode, 120microsec, 80 Hz, subthreshold for any movement or sensation, usually 3-5 volts. The stimulator will be switched off.
  Arms: B

SUMMARY:
Deep Brain Stimulation represents the golden standard for surgical treatment of Parkinson disease (PD), but it is not optimally effective for controlling every motor sign and adverse events are not so infrequent Therefore, other approaches should be considered.We identified the motor cortex as a possible candidate and therefore we propose a double-blind randomized prospective study in 20 Parkinson patients in order:

* to test the efficacy of epidural motor cortex stimulation in Parkinson disease (primary endpoint: UPDRS III at 12 months at the end of the cross-over)
* to find out optimal electrode position and optimal stimulation parameters

DETAILED DESCRIPTION:
20 Parkinsonian patients will be enrolled. After implantation of a bilateral strip electrode (Resume, Medtronic) over the motor cortex, after setting of optimal stimulation parameters, and after implantation of a neurostimulator, Medtronic, the patient will be randomly assigned to group A (Motor cortex stimulation on) or to group B ( sham stimulation) for 6 months. Randomization will be based on the output of a program based on a random number generation function that will output a 0 or 1 with a 50% chance of having a 1.

At the 6 months visit, a cross-over is scheduled: group A will receive sham stimulation and group B will receive stimulation of the motor cortex for the next 6 months. In group A, the stimulation of the motor cortex will be resumed before the end of the 6 month sham stimulation, when the clinical status of the patient will come back to the status quo ante (UPDRS score equal to baseline pre-implant score).

Both the patients and the evaluating neurologists and neuropsychologists will be blind; only the neurosurgeon will know the state of the stimulator (on or off) and the position and parameters of MCS.

At 12 months, all the patients will be programmed as stimulation on and followed up for further 18 months. At 30 months visit, the clinical evaluation will be performed in on stim-on med, on stim-off med conditions; then the stimulator will be switched off for 1 month and the clinical evaluation will be repeated in off stim-off med and off stim-on med conditions.

The primary endpoint will be the UPDRS III at 12 months (end of the cross over), and subsequently at 18 and 30 months. We will compare the clinical results with the precise site of the stimulating electrodes and we will try to correlate the clinical results with the amount of inhibition induced by motor cortex stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD as diagnosed by a neurologist - a movement disorders specialist, according to the Parkinson Disease Brain Bank criteria, with asymmetrical bradykinesia, rigidity, tremor and postural instability (at least 3 from the above)
2. Significant clinical response to Levodopa (improvement of UPDRS motor score > 20%).
3. Disease duration > 5 years
4. Advanced stage of disease:
5. UPDRS motor score in off condition >/= 40/108
6. Hoehn & Yahr stage >/= 3
7. DBS surgery not indicated or expressly refused by the patient
8. Antiparkinsonian therapy stable for at least one month prior to implant
9. Capability to give informed consent to surgery and to the study.

Exclusion Criteria:

1. Severe cognitive impairment or dementia
2. Psychiatric disturbances with the exception of mild anxiety or depression and drug-induced psychiatric symptoms (i.e. benign hallucinations)
3. History of epilepsy or documented electroencephalographic abnormalities suggesting epilepsy
4. Previous neurosurgery of the brain (DBS or lesioning of the basal ganglia, fetal tissue transplantation )
5. Lack of informed consent
6. History of drug or alcohol abuse
7. Poor general conditions increasing surgical risk or severe illness with poor prognosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
UPDRS III | 12 months - end of crossover

SECONDARY OUTCOMES:
UPDRS III | 18, 30 and 31 months
UPDRS | 6,12, 18, 30, 31 months
Parkinson's disease quality of life scale(PDQL) | 6, 12, 18, 30, 31 months
Neuropsychological and mood evaluation | 6, 12, 18, 30 months
Drug therapy | 6, 12, 18, 30, 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Cioni, MD, Principal Investigator — Università Cattolica Roma, Italy; Mario Meglio, Prof, MD, Study Chair — Università Cattolica Roma, Italy
Locations (1):
- Università Cattolica - Policlinico Gemelli - Neurochirurgia Funzionale, Roma, Italy

REFERENCES:
- [Background] Cioni B. Motor cortex stimulation for Parkinson's disease. Acta Neurochir Suppl. 2007;97(Pt 2):233-8. doi: 10.1007/978-3-211-33081-4_26. PMID 17691309
- [Background] Pagni CA, Altibrandi MG, Bentivoglio A, Caruso G, Cioni B, Fiorella C, Insola A, Lavano A, Maina R, Mazzone P, Signorelli CD, Sturiale C, Valzania F, Zeme S, Zenga F. Extradural motor cortex stimulation (EMCS) for Parkinson's disease. History and first results by the study group of the Italian neurosurgical society. Acta Neurochir Suppl. 2005;93:113-9. doi: 10.1007/3-211-27577-0_19. PMID 15986739
- [Background] Cioni B, Meglio M, Perotti V, De Bonis P, Montano N. Neurophysiological aspects of chronic motor cortex stimulation. Neurophysiol Clin. 2007 Dec;37(6):441-7. doi: 10.1016/j.neucli.2007.10.007. Epub 2007 Nov 1. PMID 18083500